CLINICAL TRIAL: NCT07384923
Title: The Effect of Vibration Devices on Pain and Discomfort During Local Anesthesia Administration in Children: A Randmized Clinical Trial.
Brief Title: The Effect of Vibration Devices on Pain and Discomfort During Local Anesthesia Administration in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Sara M.Bagher, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: KingAbdulaizU
Record Dates: First submitted 2026-01-05; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Children's Anxiety Levels; Children's Behavior; Physiological Changes (Heart Rate); Obejective Pain and Discomfort; Subjective Pain and Discomfort; Subjects' and Parents' Satisfaction; Subjects' and Parents' Future Preference
Keywords: Pain and discomfort; future preferece; satisfaction; Vibration Device
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into four groups. Those who first received maxillary buccal infiltration with the DentalVibe intraoral vibration device on the right side will be classified as group 1. Those who received it on the left side first will be classified as group 2. Meanwhile, subjects who received maxillary buccal infiltration with the Buzzy Bee® extraoral vibration device on the right side first will be classified as group 3, and those who received it on the left side first will be classified as group 4.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- The DentalVibe vibration device first on the right side then the Buzzy Bee® vibration device (Other): The DentalVibe intraoral vibration device first on the right side then the Buzzy Bee® extraoral vibration device on the left Side.
  Interventions: Device: DentalVibe intraoral vibration device; Device: Buzzy Bee® extraoral vibration device
- The DentalVibe vibration device first on the left side then the Buzzy Bee® vibration device (Other): The DentalVibe intraoral vibration device is first on the left side, then the Buzzy Bee® extraoral vibration device on the right Side.
  Interventions: Device: DentalVibe intraoral vibration device; Device: Buzzy Bee® extraoral vibration device
- The Buzzy Bee® vibration device first on the right side then the DentalVibe vibration device (Other): The Buzzy Bee® extraoral vibration device is first on the right side, then the DentalVibe intraoral vibration device on the left Side
  Interventions: Device: DentalVibe intraoral vibration device; Device: Buzzy Bee® extraoral vibration device
- The Buzzy Bee® vibration device first on the left side, then the DentalVibe vibration device (Other): The Buzzy Bee® extraoral vibration device is first on the left side, then the DentalVibe intraoral on the right side.
  Interventions: Device: DentalVibe intraoral vibration device; Device: Buzzy Bee® extraoral vibration device

INTERVENTIONS:
Device: DentalVibe intraoral vibration device — DentalVibe intraoral vibration device.
Device: Buzzy Bee® extraoral vibration device — Buzzy Bee® extraoral vibration device

SUMMARY:
This split-mouth randomized clinical trial will be conducted at the Department of Pediatric Dentistry, King Abdulaziz University Dental Hospital (KAAUDH). The inclusion criteria will include healthy, non-anxious, cooperative children aged six to 12 who require non-urgent dental treatment involving at least one pair of contralateral maxillary molars needing buccal infiltration anesthesia with no previous dental history or experience.

The children will be screened for eligibility, and a single trained dental intern will approach the parents or guardians of eligible children. Those who agree to be screened for participation in the study will be asked to sign an Arabic consent form. Before the scheduled screening appointment, children's anxiety levels will be assessed using a high score on the Abeer Children Dental Anxiety Scale (ACDAS) in the waiting area.

During the appointment, a single trained dental intern will perform the dental examination and prophylaxis, while two trained and calibrated dental interns will assess children's behavior using the Frankl Behavior Rating Scale.

Children found to be non-anxious based on their ACDAS score and cooperative or definitely cooperative based on the Frankl Behavior Rating Scale will be considered eligible for the study. Two treatment appointments will be scheduled for them, and consent and assent forms for participation in the study will be obtained.

Computer randomization will be performed to determine the treatment sequence (DentalVibe intraoral vibration device followed by Buzzy Bee® extraoral vibration device, or vice versa) and the site (right or left). Randomization will be performed before the first scheduled treatment appointment.

The subjects will be seated in the dental chair for five minutes to acclimate to the environment. To measure the physiological changes of the participating subjects, a pulse oximeter device (OxyWatch, ChoiceMMed, Hamburg, Germany) will be applied, and a trained dental intern will record the baseline heart rate (HR). During the treatment, HR will also be recorded.

The tip of the DentalVibe intraoral vibration device will be gently placed on the mucobuccal fold above the tooth to be anesthetized. In contrast, the Buzzy Bee® extraoral vibration device will be positioned externally above the buccal infiltration site.

During maxillary buccal infiltration, all subjects will be videotaped using a high-resolution camera, focusing on the face and body. Later, two trained and calibrated evaluators will independently assess the child's behavior during the procedure using the Face, Legs, Activity, Cry, Consolability Scale (FLACC) Immediately after administering anesthesia, the subjects will be positioned upright, and the same trained dental intern will introduce the face version of the Visual Analogue Scale (VAS).

Finally, after completing both procedures, the subjects will be asked about their future preference for the vibration device. Due to the study's design, both the investigator administering the maxillary buccal infiltration and the subjects will not be aware of which group they belong to.

DETAILED DESCRIPTION:
This split-mouth randomized clinical trial will be conducted at the Department of Pediatric Dentistry, King Abdulaziz University Dental Hospital (KAAUDH after obtaining ethical approval from the Research Ethics Committee of the Faculty of Dentistry, King Abdulaziz University (Reference No. 040-03-22). The study will adhere to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

The inclusion criteria will include healthy, non-anxious, cooperative children aged 6 to 12 who require non-urgent dental treatment involving at least one pair of contralateral maxillary molars, requiring buccal infiltration anesthesia, with no previous dental history or experience.

The children will be screened for eligibility by two trained dental interns during their initial regular screening appointment at KAAUDH between September and December 2025. Healthy children aged six to 12 years who require non-urgent dental treatment involving at least one pair of contralateral maxillary molars needing buccal infiltration anesthesia with no prior dental experience will be eligible for screening.

A single trained dental intern approached the parents or guardians of eligible children. Those who agree to be screened for study participation will be asked to sign an Arabic consent form. Additionally, a screening assent will be obtained from children aged seven years and older. Before the scheduled screening appointment, children's anxiety levels will be assessed using a high score on the Abeer Children Dental Anxiety Scale (ACDAS) in the waiting area. Total scores range from 13 to 39; children scoring 26 or higher are considered anxious.

During the appointment, a single trained dental intern will perform the dental examination and prophylaxis using a low-speed handpiece and a rubber cup with prophylactic paste. Two trained and calibrated dental interns will assess children's behavior during the procedure using the Frankl Behavior Rating Scale.

Children found to be non-anxious based on their ACDAS score and cooperative or definitely cooperative based on the Frankl Behavior Rating Scale will be considered eligible for the study. Two treatment appointments will be scheduled for them, and consent and assent forms for participation in the study will be obtained. Children requiring urgent dental treatment, those with active infections at the injection site, non-Arabic speakers, children with high anxiety scores in the ACDAS, or those who are uncooperative during the screening appointment will be excluded and referred to be treated by a pediatric dentist at KAAUDH.

Computer randomization will be performed to determine the treatment sequence (DentalVibe intraoral vibration device followed by Buzzy Bee® extraoral vibration device, or vice versa) and the site (right or left). Randomization will be performed before the first scheduled treatment appointment.

Subjects will be divided into four groups. Those who first received maxillary buccal infiltration with the DentalVibe intraoral vibration device on the right side will be classified as group 1. Those who received it on the left side first will be classified as group 2. Meanwhile, subjects who received maxillary buccal infiltration with the Buzzy Bee® extraoral vibration device on the right side first will be classified as group 3, and those who received it on the left side first will be classified as group 4.

The subjects will be seated in the dental chair for five minutes to acclimate to the environment. To measure the physiological changes in the participating subjects, a pulse oximeter (OxyWatch, ChoiceMMed, Hamburg, Germany) will be used, and a trained dental intern will record the baseline heart rate (HR). During the treatment, HR will also be recorded at the application of topical anesthesia, activation of the vibration device, needle insertion, and immediately after the needle is withdrawn.

Before the procedure began, the assigned device will be introduced to the subjects as a tool that causes vibrations to reduce pain and discomfort. The DentalVibe intraoral vibration device will also be presented as a tool for retracting lips and cheeks.

The mucosa at the injection site will be dried with gauze, and 20% benzocaine will be applied for 60 seconds. The tip of the DentalVibe intraoral vibration device will be gently placed on the mucobuccal fold above the tooth to be anesthetized. In contrast, the Buzzy Bee® extraoral vibration device will be positioned externally above the buccal infiltration site. The device will be operated for five seconds before needle insertion. A 30-gauge G short needle will be used. The device will remain on during buccal infiltration with 2% Mepivacaine with 1:200,000 epinephrine (Scandicaine 2% special, Septodont, UK) until five seconds after the needle is fully withdrawn. A single-trained pediatric dentist performed all the maxillary buccal infiltration administration.

During maxillary buccal infiltration, all subjects will be videotaped using a high-resolution camera, focusing on the face and body. Later, two trained and calibrated evaluators will independently assess the child's behavior during the procedure using the Face, Legs, Activity, Cry, Consolability Scale (FLACC). To ensure calibration, before the study began, the evaluators will review the behavior of 15 randomly selected children who were videotaped receiving local anesthesia using the FLACC.

Immediately after administering anesthesia, the subjects will be positioned upright, and the same trained dental intern will introduce the face version of the Visual Analogue Scale (VAS), which assesses the subject's subjective pain and discomfort. Additionally, subjects' and parents' satisfaction with each dental vibration device will be assessed.

Finally, after completing both procedures, the subjects will be asked about their future preference for the vibration device. Due to the study's design, both the investigator administering the maxillary buccal infiltration and the subjects will not be aware of which group they belong to.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children
2. Non-anxious
3. cooperative
4. Aged six to 12
5. No previous dental history or experience.

5- Who required non-urgent dental treatment involving at least one pair of contralateral maxillary molars needing buccal infiltration anesthesia

Exclusion Criteria:

1. Children requiring urgent dental treatment
2. Those with active infections at the injection site
3. Non-Arabic speakers
4. Children with high anxiety scores in the ACDAS
5. Those who were uncooperative during the screening appointment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Physiological changes (heart rate(HR)) | HR will be recorded at: 1- At baseline, onc subjects sat in the dental chair 2- At the application of topical anesthesia 3- At the activation of the vibration device 4- At needle insertion 5- Immediately after the needle is withdrawn.
  Physiological changes (HR) of the participating subjects will be measured using a pulse oximeter device (OxyWatch, ChoiceMMed, Hamburg, Germany), and a trained dental intern will record it.
The subject's subjective pain and discomfort. | Immediately after the anesthesia administration
  Visual Analogue Scale (VAS), which assesses the subject's subjective pain and discomfort. The scale is a 10-cm line that indicates the level of pain and discomfort, with zero representing no pain and 10 representing the worst possible pain.
Objective pain and discomfort | During the anesthesia administration
  Two trained and calibrated evaluators independently assessed the child's objective pain and discomfort during the procedure using the Face, Legs, Activity, Cry, Consolability Scale (FLACC). The FLACC scale ranges from 0 to 10, with 0 indicating no pain and 10 the worst possible pain.

SECONDARY OUTCOMES:
Subjects' and parents' satisfaction with each dental vibration device | Immediately after both vibration devices.
  Subjects' and parents' satisfaction with each dental vibration device will be assessed using a five-point Likert scale, where zero indicates "not satisfied at all" and 10 means "very satisfied."

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No